CLINICAL TRIAL: NCT05145491
Title: Randomized Trial Comparing Immediate Versus Deferred Surgery for Symptomatic Epiretinal Membranes
Brief Title: Randomized Trial Comparing Immediate vs. Deferred Surgery for Symptomatic ERM
Acronym: Protocol AM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRCR.net Protocol AM; UG1EY014231 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2021-12-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-09

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Vitrectomy (Active Comparator)
  Interventions: Procedure: Immediate Vitrectomy
- Deferred Vitrectomy (Other)
  Interventions: Procedure: Deferred Vitrectomy

INTERVENTIONS:
Procedure: Immediate Vitrectomy — Surgery to remove epiretinal membrane (ERM). Vitrectomy will be performed on eyes within 1 month of randomization
  Arms: Immediate Vitrectomy
Procedure: Deferred Vitrectomy — Vitrectomy may be performed only if at least one of the following criteria is met:
  1. Decrease in visual acuity ≥10 letters from baseline at a single visit presumed to be from ERM
  2. Decrease in visual acuity ≥5 letters from baseline at two consecutive visits presumed to be from ERM
     a. Visits must be at least one month apart
  3. Participant actively requests surgery due to worsening symptoms
  4. Complication requires prompt surgical intervention (e.g., macular hole, retinal detachment, non-clearing vitreous hemorrhage)
  Arms: Deferred Vitrectomy

SUMMARY:
Vitrectomy to remove an epiretinal membrane (ERM) is one of the most common procedures performed by retinal surgeons. Patients who present with significant macular changes on optical coherence tomography (OCT) but relatively good vision are often advised to defer surgery until vision declines to 20/40 or worse. However, it is unknown if delaying surgery, which allows the foveal architecture to remain compromised and potentially to deteriorate, results in worse visual acuity outcomes than if surgery is performed earlier. In addition, there is a need to better understand predictors of outcomes when surgery is performed and predictors of progression when surgery is deferred. Finally, one of the most common presenting symptoms from an ERM is distortion or metamorphopsia. There are several objective measures of metamorphopsia but none have ever been employed to evaluate ERMs in a randomized clinical trial (RCT) and their usefulness is unknown. The purposes of this study are to better understand the optimal timing of surgery to produce the best visual result, to better understand predictors of outcomes in those who undergo surgery and predictors of progression in those whose are observed, and to better characterize and evaluate the usefulness of metamorphopsia and reading speed measures.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 45 years
* E-ETDRS visual acuity 20/40 or better (≥69 letters)

  o ERM must be thought to be the primary cause of vision loss
* ERM meeting the following criteria, according to the investigator

  * ERM is not secondary to another condition
  * Symptoms of visual loss and/or distortion (in the opinion of the investigator, the ERM is contributing to the participant's symptoms); either new or worsening in the past 24 months
  * Epiretinal membrane involving or altering the central 3 mm of the macula on OCT
  * Distortion within the central subfield due to ERM on OCT
* Immediate vitrectomy not required (investigator and participant are willing to wait at least 4 weeks to see if vision remains stable without having to proceed to vitrectomy)
* No known medical problems that will be a contraindication to surgery

Key Exclusion Criteria:

* History of retinal vascular disease
* History of vitreous hemorrhage if vitreous hemorrhage is thought to have caused the ERM

  o History of vitreous hemorrhage is permitted provided the vitreous hemorrhage did not cause the ERM in the investigator's opinion
* History of inflammatory disease unless mild and completely resolved at least one year prior to randomization
* History of diabetic macular edema (DME), retinal vein occlusion (RVO), or uveitis (except mild uveitis that resolved >1 year prior to randomization)
* Prior intraocular surgery (except uncomplicated cataract extraction)
* Cataract extraction within prior 3 months
* Laser or cryosurgical retinopexy within one month of randomization
* Pneumatic retinopexy within one year of randomization
* Current untreated retinal tear or detachment

  o A previously treated retinal tear with up to one disc diameter radius of subretinal fluid is permitted
* Macular hole
* Degenerative lamellar macular hole

  o ERM foveoschisis ("tractional" lamellar hole) is permitted
* Vitreomacular traction within 1,500 microns of foveal center
* Central serous chorioretinopathy
* Nonproliferative diabetic retinopathy or worse (DR severity >20)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in visual acuity letter score from baseline to 36 months | Baseline to 36 months
  Visual acuity is measured as a continuous integer letter score from 0 to 100, with higher numbers indicating better visual acuity. A letter score of 85 is approximately 20/20 and a letter score of 70 is approximately 20/40, the legal unrestricted driving limit in most states. A 5-letter change for an individual is approximately equal to a 1-line change on a vision chart.

CONTACTS AND LOCATIONS:
Locations (46):
- United States (45):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Kent W. Small, MD, AMC, Glendale, California
  - Salehi Retina Institute Inc., Huntington Beach, California
  - Loma Linda University, Loma Linda, California
  - Retina Vitreous Associates, Northern California Retina Vitreous Assoc Medical Group, Inc., Mountain View, California
  - East Bay Retina Consultants, Inc., Oakland, California
  - Regents of the University of California, Davis, DBA University of California, Davis, Sacramento, California
  - Macula Retina Vitreous Institute, Torrance, California
  - Florida Retina Institute, James A. Staman, MD, PA- Jacksonville, Jacksonville, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - SEASHORE RETINA LLC DBA Retina Specialists of Tampa, Wesley Chapel, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Illinois Retina Associates SC - Oak Park Site, Oak Park, Illinois
  - Raj K. Maturi, M.D., P.C., Indianapolis, Indiana
  - Mid-America Retina Consultants, P.A., Overland Park, Kansas
  - University of Kansas Medical Center Research Institute, Inc., Prairie Village, Kansas
  - Joseph E. Humble and Raymond Haik PTRS DBA Eye Assoc of Northeast Louisiana, West Monroe, Louisiana
  - Elman Retina Group, P.A., Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Retina Associates of Michigan, Grand Blanc, Michigan
  - The Curators of the University of Missouri, Columbia, Missouri
  - Retina Research Institute, LLC, St Louis, Missouri
  - Retina-Vitreous Surgeons of Central NY, PC, Liverpool, New York
  - Retina Associates of Western NY, P.C., Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Retina Vitreous Center, Edmond, Oklahoma
  - Verum Research LLC, Eugene, Oregon
  - Cascade Medical Research Institute, LLC, Springfield, Oregon
  - Retina-Vitreous Consultants, Inc., Monroeville, Pennsylvania
  - The Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pittsburg Clinical Trial Consortium, Sewickley, Pennsylvania
  - Hilton Head Retina Institute, Hilton Head Island, South Carolina
  - Ophthalmology Ltd., Sioux Falls, South Dakota
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Austin Research Center for Retina, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Baylor College of Medicine, Baylor Eye Physicians and Surgeons, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Spokane Eye Clinical Research, PLLC, Spokane, Washington
- South Tyneside and Sunderland NHS Trust, Sunderland, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No